CLINICAL TRIAL: NCT00793143
Title: A Randomized Prospective Three-center Study: Laparoscopic Gastric Bypass vs. Laparoscopic Sleeve Gastrectomy in the Treatment of Morbid Obesity
Brief Title: Laparoscopic Gastric Bypass Versus Sleeve Gastrectomy to Treat Morbid Obesity
Acronym: SLEEVEPASS
Status: Completed | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Collaborators: Vaasa Central Hospital, Vaasa, Finland (Other); Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Paulina Salminen, MD, PhD, Turku University Hospital
Other Study IDs: SLEEVEPASS
Record Dates: First submitted 2008-11-17; First posted 2008-11-19 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Morbid Obesity
Keywords: morbid obesity; laparoscopic sleeve gastrectomy; LSG; laparoscopic gastric bypass; LGB; comorbidities; diabetes; excessive weight loss; weight loss
MeSH Terms: conditions — Obesity, Morbid; Diabetes Mellitus; Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Sleeve
- Bypass

SUMMARY:
Bariatric surgery in the treatment of morbid obesity is associated with long-term weight-loss and decreased overall mortality. Long-term results have been reported for laparoscopic gastric bypass procedures but the long-term results of laparoscopic sleeve gastrectomy are yet unavailable. As sleeve gastrectomy is a rapid and less traumatic procedure with good short-term results of weight loss and resolution of comorbidities, the investigators initiated a prospective randomized two-center study comparing laparoscopic sleeve gastrectomy (LSG)with laparoscopic gastric bypass (LGB) in the treatment of morbid obesity. Study hypothesis: As sleeve gastrectomy is less traumatic, easier and faster to perform compared with gastric bypass,LSG could become the procedure of choice to treat morbid obesity if the long-term results of weight loss and resolution of comorbidities are comparable with laparoscopic gastric bypass.

DETAILED DESCRIPTION:
In addition to comparing the outcomes between sleeve gastrectomy and gastric bypass, the study project includes a PET trial conducted in Turku. The objectives of this PET study are to measure effect of obesity on food-stimuli mediated brain activation response and on hormones affecting both feeding and energy balance. In the second part the same variables are studied after bariatric surgery: either laparoscopic sleeve gastrectomy or Roux-en-Y gastric bypass. In addition the effect of weight loss due to bariatric surgery on glucose uptake and free fatty acid metabolism is measured. The objective is also to study whether less invasive sleeve gastrectomy is as beneficial in terms of weight loss and co-morbid diseases as more invasive Roux-en-Y gastric bypass and to compare the risk factors between these two surgical procedures. Regional glucose uptake and free fatty acid uptake in myocardium, skeletal muscle, subcutaneous fat, visceral fat, pancreas, liver and brain are studied with PET at baseline before bariatric surgery and post-operatively on the 3rd month. Changes in body fat distribution, in ectopic fat and fat content of key organs are investigated with magnetic resonance imaging (MRI) and magnetic resonance spectroscopy (MRS). Brain reward system response to food stimuli is assessed using functional MRI (fMRI) and white and grey matter volumes using diffusion tensor imaging (DTI).

The study consists of 80 morbidly obese adults, BMI ≥ 40 kg/m2 or if there is additional risk factor BMI ≥ 35 kg/m2. From these subjects, 40 are further studied with positron emission tomography (PET) and magnetic resonance imaging (MRI). In addition functional MRI (fMRI) will be performed for 40 subjects. For fMRI, a control group is recruited consisting of 20 lean and healthy subjects. Subjects are physically examined and anthropometric data are measured along with blood sampling.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 40 or BMI > 35 with a comorbidity associated with obesity
* Age 18 - 60 years
* Failed prior effective and controlled conservative treatments of morbid obesity

Exclusion Criteria:

* BMI > 60
* Difficult psychiatric conditions or lack of co-operation
* Difficult eating disorder (binge eating, bulimia etc.)
* Alcohol abuse
* Gastric ulcer

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients rederred to three tertiary referral hospitals (Turku University Central Hospital, Vaasa Central Hospital and Peijas Hospital)for treatment of morbid obesity
Sampling Method: Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2008-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Excessive weight loss | 3,6,12,18 months, 2,3,5,7,10,15 years

SECONDARY OUTCOMES:
Resolution of comorbidities | 3,6,12,18 months, 2,3,5,7,10,15 years
Mortality | 0 - 15 years
Morbidity | 0 - 15 years
QOL (15D and BAROS) | 3,6,12,18 months, 2,3,5,7,10,15 years

CONTACTS AND LOCATIONS:
Overall Officials: Paulina Salminen, MD, PhD, Principal Investigator — Turku Univeristy Central Hospital; Jari Ovaska, Md, PhD, Principal Investigator — University of Turku; Mikael Victorzon, MD, PhD, Principal Investigator — Vaasa Central Hospital, Vaasa, Finland
Locations (4):
- Finland (4):
  - Helsinki University Hospital, Helsinki
  - Department of Surgery, Turku University Central Hospital, Turku
  - Turku University Hospital, PET-center, Turku
  - Vaasa Central Hospital, Vaasa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dadson P, Honka MJ, Suomi T, Rokka A, Kauhanen S, Salminen P, Helmio M, James P, Elo LL, Olkkonen VM, Nuutila P. Characterization of Visceral Adipose Tissue Proteome Reveals Metabolic Changes and Inflammatory Signatures in Severe Obesity. Obesity (Silver Spring). 2026 Jan;34(1):127-137. doi: 10.1002/oby.70041. Epub 2025 Oct 12. PMID 41077621
- [Derived] Dadson P, Rebelos E, Jaakkola MK, Monfort-Pires M, Ojala R, Honka H, Kalliokoski KK, Klen R, Nuutila P, Ivaska KK. Differential associations of subcutaneous and visceral fat with bone turnover markers: A study on bariatric surgery patients with severe obesity and individuals without obesity. Int J Obes (Lond). 2025 Dec;49(12):2494-2502. doi: 10.1038/s41366-025-01888-1. Epub 2025 Aug 26. PMID 40854969
- [Derived] Saarinen I, Strandberg M, Hurme S, Helmio M, Gronroos S, Juuti A, Juusela R, Nuutila P, Salminen P. Nutritional deficiencies after sleeve gastrectomy and Roux-en-Y gastric bypass at 10 years: secondary analysis of the SLEEVEPASS randomized clinical trial. Br J Surg. 2025 Jul 3;112(7):znaf132. doi: 10.1093/bjs/znaf132. PMID 40613787
- [Derived] Dadson P, Honka MJ, Suomi T, Haridas PAN, Rokka A, Palani S, Goltseva E, Wang N, Roivainen A, Salminen P, James P, Olkkonen VM, Elo LL, Nuutila P. Proteomic profiling reveals alterations in metabolic and cellular pathways in severe obesity and following metabolic bariatric surgery. Am J Physiol Endocrinol Metab. 2025 Mar 1;328(3):E311-E324. doi: 10.1152/ajpendo.00220.2024. Epub 2025 Jan 17. PMID 39819027
- [Derived] Saarinen I, Strandberg M, Hurme S, Gronroos S, Juuti A, Helmio M, Salminen P. Association of High-Sensitivity C-Reactive Protein (hs-CRP) with Weight Loss After Sleeve Gastrectomy and Roux-en-Y Gastric Bypass at 10 Years: A Secondary Analysis of the SLEEVEPASS Randomized Clinical Trial. Obes Surg. 2024 Dec;34(12):4378-4384. doi: 10.1007/s11695-024-07567-w. Epub 2024 Nov 7. PMID 39509008
- [Derived] Peterli R, Hurme S, Bueter M, Gronroos S, Helmio M, Salminen P. Standardized Assessment of Metabolic Bariatric Surgery Outcomes: Secondary Analysis of 2 Randomized Clinical Trials. JAMA Surg. 2024 Mar 1;159(3):306-314. doi: 10.1001/jamasurg.2023.6254. PMID 38055284
- [Derived] Saux P, Bauvin P, Raverdy V, Teigny J, Verkindt H, Soumphonphakdy T, Debert M, Jacobs A, Jacobs D, Monpellier V, Lee PC, Lim CH, Andersson-Assarsson JC, Carlsson L, Svensson PA, Galtier F, Dezfoulian G, Moldovanu M, Andrieux S, Couster J, Lepage M, Lembo E, Verrastro O, Robert M, Salminen P, Mingrone G, Peterli R, Cohen RV, Zerrweck C, Nocca D, Le Roux CW, Caiazzo R, Preux P, Pattou F. Development and validation of an interpretable machine learning-based calculator for predicting 5-year weight trajectories after bariatric surgery: a multinational retrospective cohort SOPHIA study. Lancet Digit Health. 2023 Oct;5(10):e692-e702. doi: 10.1016/S2589-7500(23)00135-8. Epub 2023 Aug 29. PMID 37652841
- [Derived] Salminen P, Gronroos S, Helmio M, Hurme S, Juuti A, Juusela R, Peromaa-Haavisto P, Leivonen M, Nuutila P, Ovaska J. Effect of Laparoscopic Sleeve Gastrectomy vs Roux-en-Y Gastric Bypass on Weight Loss, Comorbidities, and Reflux at 10 Years in Adult Patients With Obesity: The SLEEVEPASS Randomized Clinical Trial. JAMA Surg. 2022 Aug 1;157(8):656-666. doi: 10.1001/jamasurg.2022.2229. PMID 35731535
- [Derived] Gronroos S, Helmio M, Juuti A, Tiusanen R, Hurme S, Loyttyniemi E, Ovaska J, Leivonen M, Peromaa-Haavisto P, Maklin S, Sintonen H, Sammalkorpi H, Nuutila P, Salminen P. Effect of Laparoscopic Sleeve Gastrectomy vs Roux-en-Y Gastric Bypass on Weight Loss and Quality of Life at 7 Years in Patients With Morbid Obesity: The SLEEVEPASS Randomized Clinical Trial. JAMA Surg. 2021 Feb 1;156(2):137-146. doi: 10.1001/jamasurg.2020.5666. PMID 33295955
- [Derived] Pham TT, Ivaska KK, Hannukainen JC, Virtanen KA, Lidell ME, Enerback S, Makela K, Parkkola R, Piirola S, Oikonen V, Nuutila P, Kiviranta R. Human Bone Marrow Adipose Tissue is a Metabolically Active and Insulin-Sensitive Distinct Fat Depot. J Clin Endocrinol Metab. 2020 Jul 1;105(7):2300-10. doi: 10.1210/clinem/dgaa216. PMID 32311037
- [Derived] Savolainen AM, Karmi A, Immonen H, Soinio M, Saunavaara V, Pham T, Salminen P, Helmio M, Ovaska J, Loyttyniemi E, Heiskanen MA, Lehtimaki T, Mari A, Nuutila P, Hannukainen JC. Physical Activity Associates with Muscle Insulin Sensitivity Postbariatric Surgery. Med Sci Sports Exerc. 2019 Feb;51(2):278-287. doi: 10.1249/MSS.0000000000001778. PMID 30247434
- [Derived] Salminen P, Helmio M, Ovaska J, Juuti A, Leivonen M, Peromaa-Haavisto P, Hurme S, Soinio M, Nuutila P, Victorzon M. Effect of Laparoscopic Sleeve Gastrectomy vs Laparoscopic Roux-en-Y Gastric Bypass on Weight Loss at 5 Years Among Patients With Morbid Obesity: The SLEEVEPASS Randomized Clinical Trial. JAMA. 2018 Jan 16;319(3):241-254. doi: 10.1001/jama.2017.20313. PMID 29340676
- [Derived] Honka H, Hannukainen JC, Tarkia M, Karlsson H, Saunavaara V, Salminen P, Soinio M, Mikkola K, Kudomi N, Oikonen V, Haaparanta-Solin M, Roivainen A, Parkkola R, Iozzo P, Nuutila P. Pancreatic metabolism, blood flow, and beta-cell function in obese humans. J Clin Endocrinol Metab. 2014 Jun;99(6):E981-90. doi: 10.1210/jc.2013-4369. Epub 2014 Feb 14. PMID 24527718
- [Derived] Immonen H, Hannukainen JC, Iozzo P, Soinio M, Salminen P, Saunavaara V, Borra R, Parkkola R, Mari A, Lehtimaki T, Pham T, Laine J, Karja V, Pihlajamaki J, Nelimarkka L, Nuutila P. Effect of bariatric surgery on liver glucose metabolism in morbidly obese diabetic and non-diabetic patients. J Hepatol. 2014 Feb;60(2):377-83. doi: 10.1016/j.jhep.2013.09.012. Epub 2013 Sep 20. PMID 24060855
- [Derived] Tuulari JJ, Karlsson HK, Hirvonen J, Hannukainen JC, Bucci M, Helmio M, Ovaska J, Soinio M, Salminen P, Savisto N, Nummenmaa L, Nuutila P. Weight loss after bariatric surgery reverses insulin-induced increases in brain glucose metabolism of the morbidly obese. Diabetes. 2013 Aug;62(8):2747-51. doi: 10.2337/db12-1460. Epub 2013 Mar 14. PMID 23493575